CLINICAL TRIAL: NCT06821269
Title: Functional Recovery After Total Knee Arthroplasty
Status: Recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Kenneth Urish, Associate Professor, University of Pittsburgh
Other Study IDs: STUDY23060125
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Arthritis Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Manual Revision TKA: These patients underwent revision TKA done manually
  Interventions: Procedure: Manual revision total knee arthroplasty
- Robotic-assisted Revision TKA: These patients underwent revision TKA with robotic-assistance
  Interventions: Procedure: Robotic assisted revision total knee arthroplasty
- Manual Primary TKA: These patients received primary TKAs done manually
  Interventions: Procedure: Manual total knee arthroplasty
- Robotic-assisted Primary TKA: These patients received primary TKAs with robotic-assistance
  Interventions: Procedure: Robotic assisted total knee arthroplasty

INTERVENTIONS:
Procedure: Robotic assisted total knee arthroplasty — Total knee arthroplasty with robotic assisatance
  Groups: Robotic-assisted Primary TKA
Procedure: Manual total knee arthroplasty — Total knee arthroplasty without robotic assistance
  Groups: Manual Primary TKA
Procedure: Robotic assisted revision total knee arthroplasty — Revision total knee arthroplasty with robotic assistance
  Groups: Robotic-assisted Revision TKA
Procedure: Manual revision total knee arthroplasty — Revision total knee arthroplasty without robotic assistance
  Groups: Manual Revision TKA

SUMMARY:
The goal of this observational study is to learn about patients' recoveries after receiving total knee arthroplasty (TKA). The main questions it aims to answer are:

Does robotic-assisted TKA have improved perceived recovery when compared to conventional TKA? Does robotic-assisted TKA lead to improved functional recovery when compared to conventional TKA?

Researchers will compare if robotic-assisted versus conventional procedures lead to different recovery speeds.

Participants will answer questionnaires and undergo physical therapy testing before and at several timepoints after their procedure.

DETAILED DESCRIPTION:
The choice to perform robotic assisted vs manual total knee arthroplasties (TKA) depends on many factors, including but not limited to surgeon training, resource availability, and patient-specific considerations. Recent studies comparing patient outcomes after robotic-assisted and manual total knee arthroplasties have shown mixed results. These studies often focus on future complication rates, radiographic outcomes, or patient reported outcomes between manual and robotic-assisted TKA. Hence, there has been little focus on improvements in functional outcomes after TKA. Combining functional test results, patient reported outcomes, kinematic studies, and data from wearable devices will allow for a comprehensive timeline of recovery speed after either robotic-assisted or manual TKA.

The overall aim of this proposed study is to quantify functional and PROM at specific timepoints in patients after robotic-assisted or manual total knee arthroplasty (TKA).

The questions are:

1. Do robotic-assisted revision TKAs have improved functional and perceived recovery when compared to manual revision TKAs?
2. Do robotic-assisted primary TKAs have improved functional and perceived recovery when compared to manual primary TKAs?
3. Do robotic-assisted revision TKAs have similar functional and perceived recovery as robotic-assisted primary TKAs?

For questions 1 and 2, we hypothesize that robotic-assisted revision or primary TKAs will have improved recovery when compared to manual TKAs.

For question 3, we hypothesize that robotic-assisted revision TKA will have similar recovery to primary robotic-assisted TKA.

Patients who are candidates for revision or primary TKA will be recruited within the Department of Orthopaedic Surgery. All subjects will participate in 6 evaluation sessions: anytime pre-operatively (baseline) and 2 weeks, 6 weeks, 3 months, 6 months, and 1 year post surgery. Testing sessions will be approximately 1 hour long and will take place at the Physical Therapy Clinical and Translational Research Center (PT-CTRC).

At the time of enrollment, subjects will sign the informed consent in the presence of a study investigator. The research coordinator will collect data on demographics, medical history, and biomedical information. Note: Subjects who do not sign the consent form cannot participate in the study.

At each evaluation, patients will then be given time to complete the following patient reported outcome questionnaires: Forgotten Joint, Promis 29, Koos, SF 36. The physical therapist will then lead the patient through a series of functional measurement tests: Timed Up and Go (TUG), 4m and 10m walking speed test, sit/stand, Star Excursion Balance Test (SEBT), 2-minute walk, stair climb test (SCT), Single Leg Stance (SLS), and Y Balance Test (YBT). Videos may be taken to record progress.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for TKA
* Speak English / understand study instructions--this is necessary to reliably complete the study questionnaires and understand study instructions which are not validated in other languages
* Have medical clearance from PCP, PI, or co-Investigator to participate in the study
* Willing to comply with all study procedures and be available for the duration of the study

Exclusion Criteria:

* 2+ falls in the past year
* Unable to ambulate 100 ft without assistive device or rest period
* Acute illness
* Have a history of cardiovascular disease or hypertension not controlled by medication
* Severe visual impairment
* Lower-extremity amputation
* Neurological, muscular, systemic, or connective tissue disorder affecting the function of the lower extremities
* Pregnant
* Terminal illness
* Plans to have another joint replacement during study period
* Plans to relocate from immediate area during study period

Ages: 40 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients who are candidates for primary or revision total knee arthroplasty.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Timed Up and Go (TUG) | anytime pre-operatively (baseline) and 2 weeks, 6 weeks, 3 months, 6 months, and 1 year post surgery
  TUG requires the patient to sit in a chair, stand, walk to a line 3m away, turn, walk back to the chair, and sit again
4m and 10m Walking Speed Test | anytime pre-operatively (baseline) and 2 weeks, 6 weeks, 3 months, 6 months, and 1 year post surgery
2-minute Walk | anytime pre-operatively (baseline) and 2 weeks, 6 weeks, 3 months, 6 months, and 1 year post surgery
Stair Climb Test | anytime pre-operatively (baseline) and 2 weeks, 6 weeks, 3 months, 6 months, and 1 year post surgery
Y Balance Test | anytime pre-operatively (baseline) and 2 weeks, 6 weeks, 3 months, 6 months, and 1 year post surgery
  The YBT requires the person to balance on one leg whilst simultaneously reaching as far as possible with the other leg in three separate directions: anterior, posterolateral, and posteromedial

SECONDARY OUTCOMES:
Forgotten Joint Score | anytime pre-operatively (baseline) and 2 weeks, 6 weeks, 3 months, 6 months, and 1 year post surgery
  The Forgotten Joint Score (FJS) is a 12-question patient-reported outcomes measure created to measure a patient's awareness of their artificial joint.
Promis | anytime pre-operatively (baseline) and 2 weeks, 6 weeks, 3 months, 6 months, and 1 year post surgery
  PROMIS stands for Patient Reported Outcomes Measurement Information System, which is a system of highly reliable, precise measures of patient-reported health status for physical, mental, and social well-being
SF36 | anytime pre-operatively (baseline) and 2 weeks, 6 weeks, 3 months, 6 months, and 1 year post surgery
  The Short Form 36 Health Survey Questionnaire (SF-36) is used to indicate the health status of particular populations, to help with service planning and to measure the impact of clinical and social interventions.
KOOS | anytime pre-operatively (baseline) and 2 weeks, 6 weeks, 3 months, 6 months, and 1 year post surgery
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) is a 42-item questionnaire that helps patients and therapists assess knee injury outcomes over time

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Urish, MD PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No